CLINICAL TRIAL: NCT00960063
Title: A Phase 1/1B Dose-Escalation Study to Determine the Safety and Tolerability of SCH 717454 Administered in Combination With Chemotherapy in Pediatric Subjects With Advanced Solid Tumors (Protocol No. 05883)
Brief Title: A Study of Robatumumab (SCH 717454, MK-7454) in Combination With Different Treatment Regimens in Pediatric Participants With Advanced Solid Tumors (P05883, MK-7454-006)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated for business reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05883; MK-7454-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Neoplasms; Solid Tumors; Bone Cancer; Kidney Tumor; Neuroblastoma
MeSH Terms: conditions — Neoplasms; Bone Neoplasms; Carcinoma, Renal Cell; Neuroblastoma | interventions — Temozolomide; Vincristine; Ifosfamide; Irinotecan; robatumumab; Doxorubicin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Temozolomide+Irinotecan+Robatumumab (Experimental): Participants receive temozolomide 100 mg/m^2/day intravenously (IV) on Days 1-5 PLUS irinotecan 10 mg/m^2/day IV on Days 1-5 and Days 8-12 PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 3-week cycle.
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Biological: Robatumumab
- Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab (Experimental): Participants receive vincristine 2 mg/m^2 (maximum 2 mg) IV on Day 1 PLUS cyclophosphamide 1200 mg/m^2 IV on Day 1 PLUS doxorubicin hydrochloride 75 mg/m^2 IV continuously over 48 hours PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 3-week cycle.
  Interventions: Drug: Vincristine; Biological: Robatumumab; Drug: Doxorubicin; Drug: Cyclophosphamide
- Ifosfamide+Etoposide+Robatumumab (Experimental): Participants receive ifosfamide 1800 mg/m^2 per day IV PLUS etoposide 100 mg/m^2 per day IV on Days 1-5 PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 3-week cycle.
  Interventions: Drug: Ifosfamide; Biological: Robatumumab; Drug: Etoposide

INTERVENTIONS:
Drug: Temozolomide
  Arms: Temozolomide+Irinotecan+Robatumumab
Drug: Vincristine
  Arms: Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab
Drug: Ifosfamide
  Arms: Ifosfamide+Etoposide+Robatumumab
Drug: Irinotecan
  Arms: Temozolomide+Irinotecan+Robatumumab
Biological: Robatumumab
Drug: Doxorubicin
  Arms: Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab
Drug: Cyclophosphamide
  Arms: Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab
Drug: Etoposide
  Arms: Ifosfamide+Etoposide+Robatumumab

SUMMARY:
This is a Phase 1/1B, non-randomized, open-label, dose-escalation study of robatumumab (SCH 717454, MK-7454) administered in combination with chemotherapy in pediatric participants with solid tumors, to be conducted in conformance with Good Clinical Practices. This study will evaluate the safety, tolerability and dose-finding of robatumumab when administered in combination with temozolomide and irinotecan (Arm A); or cyclophosphamide, doxorubicin, and vincristine (Arm B), or ifosfamide and etoposide (Arm C).

The primary study hypothesis is that robatumumab can be safely administered in combination with chemotherapy regimens in pediatric participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must be <= 21 years of age (older participants may be allowed on study on a case-by-case basis); may be of either sex, and of any race/ethnicity.
* Must have histologic confirmation of the advanced solid tumor, except for brainstem tumors.
* Must have Karnofsky performance score of >=50 (if participant is >16 years of age) or a Lansky score of >50 (if participant is <=16 years of age).
* Must have adequate organ function during Screening.
* Must be able to adhere to dose and visit schedules.

Exclusion Criteria:

* Must not have a history of another malignancy.
* Must not have uncontrolled diabetes mellitus.
* Must not have persistent, unresolved common terminology criteria for adverse events (CTCAE) Grade >=2 drug-related toxicity associated with previous treatment.
* Must not have known hypersensitivity to other antibodies, or any accompanying excipients associated with these medications.
* If female, must not be breast-feeding, pregnant, intending to become pregnant, or have a positive pregnancy test at Screening.
* Must not be known to have human immunodeficiency virus (HIV) infection or known HIV-related malignancy.
* Must not be known to have active Hepatitis B, or Hepatitis C.
* Must not have any serious or uncontrolled infection.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2009-11-11 (Actual); Primary Completion 2010-12-22 (Actual); Study Completion 2010-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05883&kw=P05883&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Started | 1 | 0 | 3
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Progression of Disease | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Temozolomide+Irinotecan+Robatumumab: Participants receive temozolomide 100 mg/m^2/day IV on Days 1-5 PLUS irinotecan 10 mg/m^2/day IV on Days 1-5 and Days 8-12 PLUS robatumumab 10 mg/kg or 20 mg/kg IV on Day 1 of each 3-week cycle.
- Total: Total of all reporting groups
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab | Total
Number analyzed (Participants) | 1 | 0 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.0 (0.0) |  | 8.3 (4.5) | 12.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0 | 0
  Male | 1 |  | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose-limiting toxicity was defined by the following adverse events (AEs) that were considered possibly or probably related to either robatumumab or to its interaction with the chemotherapy regimen assigned: neutropenia (Grade 4 for >1 week that did not resolve prior to Day 1 of the next cycle; Grade 3-4 neutropenia with Grade ≥2 fever lasting 3 days; neutropenic infection; failure to recover to study entry/eligibility criteria laboratory requirement levels that resulted in a delay of 14 days between treatment cycles), thrombocytopenia (Grade 4 for >1 week that did not resolve prior to Day 1 of the next cycle; Grade 3-4 requiring a platelet transfusion on 2 separate days within a cycle) or all other AEs (Grade ≥3 [any duration] not ameliorable by supportive or symptomatic measures). The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version 4.0) was to be used to grade AEs.
Time Frame: Up to ~30 days after last dose of study drug (Up to ~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy.
Measure: Number; unit: Participants
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 1 | 0 | 3
Participants | 1 |  | 3

2. Secondary Outcome: Best Overall Response Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs were to be identified as target lesions. Data were to be collected at Screening, every 6 weeks and at 30 days after the final dose of robatumumab or the standard treatment assigned (whichever was last). The best overall response was to be the best response recorded from the start of the treatment until disease progression/recurrence. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >30% decrease in the sum of the longest diameter (LD) of target lesions; Progressive Disease (PD): >20% increase in the sum of the LD of target lesions or the appearance of one or more new lesions; or Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Screening, every 6 weeks and at ~30 days after last dose of study drug (Up to ~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy.
Measure: Number; unit: Participants
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 1 | 0 | 3
Participants
  Complete Response (CR) | 0 |  | 0
  Partial Response (PR) | 1 |  | 2
  Stable Disease (SD) | 0 |  | 0
  Progressive Disease (PD) | 0 |  | 1

3. Secondary Outcome: Maximum Observed Concentration (Cmax) of Robatumumab
Description: Cmax was defined as the maximum observed serum concentration of robatumumab when administered in combination with other treatments. Blood samples for analysis of robatumumab pharmacokinetics (PK) were to be obtained at Cycles 1 and 2 at the following time points: predose, immediately post-infusion, and at 3, 6, 24, 48, 168, 336, and 504 hours post the start time of infusion. For all odd-numbered cycles (Cycle 3 and on) samples were to be obtained at each of the following two time points: predose and immediately postdose of robatumumab. Additionally, PK samples were to be obtained at the Post Study Visits 1 (30 days after last dose of robatumumab or standard treatment and 2 (approximately 4 months after last dose of robatumumab or standard treatment).
Time Frame: Cycles 1 & 2: pre- and post-infusion, and at 3, 6, 24, 48, 168, 336, and 504 hours post start of infusion; then pre-and post-dose in odd-numbered cycles, and Post Study Visits 1 and 2
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for Cmax were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Plasma Level of Insulin-like Growth Factor-I (IGF-I)
Description: IGF-I is produced largely by the liver in response to growth hormone from the hypothalamic-pituitary axis. The IGF ligands can promote neoplastic events (cancer growth) through a number of different mechanisms. Robatumumab inhibits IGF ligand binding, IGF-stimulated receptor phosphorylation and human tumor cell proliferation. Plasma levels of IGF-I were to be analyzed on Day 1 of Cycles 1, 2, 3, 5, and approximately 30 days after the final dose of robatumumab or the standard treatment assigned (whichever was last).
Time Frame: On Day 1 of Cycles 1, 2, 3 and 5, and ~30 days after last dose of study drug (Up to~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for IGF-I were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Who Developed Anti-robatumumab Antibodies
Description: The incidence of anti-robatumumab antibodies was to be assessed. Only participants who had a negative pre-treatment sample and a post-treatment sample were considered to be evaluable. If a participant had a single sample considered positive in the anti-robatumumab antibody assay (with the exception of pre-treatment positive participants), then they would be counted as positive in the immunogenicity assessment.
Time Frame: Prior to 1st and 8th doses of robatumumab, ~30 days after last dose of study drug, and 4 months after last dose of study drug (Up to ~13.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy and had a negative pre-treatment sample and a post-treatment sample.
Measure: Number; unit: Participants
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 1 | 0 | 2
Participants | 0 |  | 0

6. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Robatumumab
Description: Tmax was defined as time of Cmax of robatumumab when administered in combination with other treatments. Blood samples for analysis of robatumumab PK were to be obtained at Cycles 1 and 2 at the following time points: predose, immediately post-infusion, and at 3, 6, 24, 48, 168, 336, and 504 hours post the start time of infusion. For all odd-numbered cycles (Cycle 3 and on) samples were to be obtained at each of the following two time points: predose and immediately postdose of robatumumab. Additionally, PK samples were to be obtained at the Post Study Visits 1 (30 days after last dose of robatumumab or standard treatment and 2 (approximately 4 months after last dose of robatumumab or standard treatment).
Time Frame: as for outcome 3
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for Tmax were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Area Under the Curve at the Time of Final Quantifiable Sample (AUCtf) for Robatumumab
Description: AUCtf for robatumumab was defined as the area under the curve at the time of the final quantifiable sample of robatumumab. Blood samples for analysis of robatumumab PK were to be obtained at Cycles 1 and 2 at the following time points: predose, immediately post-infusion, and at 3, 6, 24, 48, 168, 336, and 504 hours post the start time of infusion. For all odd-numbered cycles (Cycle 3 and on) samples were to be obtained at each of the following two time points: predose and immediately postdose of robatumumab. Additionally, PK samples were to be obtained at the Post Study Visits 1 (30 days after last dose of robatumumab or standard treatment and 2 (approximately 4 months after last dose of robatumumab or standard treatment).
Time Frame: as for outcome 3
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for AUCtf were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Area Under the Curve During a Dosing Interval τ (AUCτ) for Robatumumab
Description: AUCτ was defined as the area under the plasma concentration-time curve during a dosage interval (τ). Blood samples for analysis of robatumumab PK were to be obtained at Cycles 1 and 2 at the following time points: predose, immediately post-infusion, and at 3, 6, 24, 48, 168, 336, and 504 hours post the start time of infusion. For all odd-numbered cycles (Cycle 3 and on) samples were to be obtained at each of the following two time points: predose and immediately postdose of robatumumab. Additionally, PK samples were to be obtained at the Post Study Visits 1 (30 days after last dose of robatumumab or standard treatment and 2 (approximately 4 months after last dose of robatumumab or standard treatment).
Time Frame: as for outcome 3
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for AUCτ were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Plasma Level of Insulin-like Growth Factor-2 (IGF-II)
Description: IGF-II is generally produced locally in response to growth hormone from the hypothalamic-pituitary axis. The IGF ligands can promote neoplastic events (cancer growth) through a number of different mechanisms. Robatumumab inhibits IGF ligand binding, IGF-stimulated receptor phosphorylation and human tumor cell proliferation. Plasma levels of IGF-II were to be analyzed on Day 1 of Cycles 1, 2, 3, 5, and approximately 30 days after the final dose of robatumumab or the standard treatment assigned (whichever was last).
Time Frame: On Day 1 of Cycles 1, 2, 3 and 5, and ~30 days after last dose of study drug (Up to~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for IGF-II were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Plasma Level of Insulin-like Growth Factor Binding Protein-2 (IGFBP-2)
Description: The IGFBP-2 protein is secreted into the bloodstream where it binds to IGF-I and IGF-II. High expression levels of this protein promote the growth of several types of tumors and may be predictive of the chances of recovery of the participant. Robatumumab inhibits expression of this protein. Plasma levels of IGFBP-2 were to be analyzed on Day 1 of Cycles 1, 2, 3, 5, and approximately 30 days after the final dose of robatumumab or the standard treatment assigned (whichever was last).
Time Frame: On Day 1 of Cycles 1, 2, 3 and 5, and ~30 days after last dose of study drug (Up to~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for IGFBP-2 were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Plasma Level of Insulin-like Growth Factor Binding Protein-3 (IGFBP-3)
Description: The IGFBP-3 protein is secreted into the bloodstream where it binds to IGF-I and IGF-II. High expression levels of this protein promote the growth of several types of tumors and may be predictive of the chances of recovery of the participant. Robatumumab inhibits expression of this protein. Plasma levels of IGFBP-3 were to be analyzed on Day 1 of Cycles 1, 2, 3, 5, and approximately 30 days after the final dose of robatumumab or the standard treatment assigned (whichever was last).
Time Frame: On Day 1 of Cycles 1, 2, 3 and 5, and ~30 days after last dose of study drug (Up to~10.3 months)
Population: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy. Individual data were collected, but, due to study termination and small numbers of participants, summary data for IGFBP-3 were not produced.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to ~10.3 months)
Description: All Treated Set was defined as all participants who received ≥1 dose of robatumumab or chemotherapy.
Arm/Group | Temozolomide+Irinotecan+Robatumumab | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab | Ifosfamide+Etoposide+Robatumumab
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide+Irinotecan+Robatumumab (N=1) | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab (N=0) | Ifosfamide+Etoposide+Robatumumab (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide+Irinotecan+Robatumumab (N=1) | Vincristine+Doxorubicin+Cyclophosphamide+Robatumumab (N=0) | Ifosfamide+Etoposide+Robatumumab (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (18)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (12)
Thromobocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (13)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (6)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (8)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.